CLINICAL TRIAL: NCT05669521
Title: A Phase 2a, Multi-centre, Placebo Controlled, Randomized, Assessor Blind Study of Bolus 5-fluorouracil and Infused Leucovorin Plus Either Infused TK-90 for Parenteral Use or Infused TK-90 Placebo Administered Weekly for 6 Consecutive Weeks to Patients With Colorectal Cancer.
Brief Title: Phase 2a Study to Evaluate Suppression of 5-Fluorouracil -Induced Mucositis by TK112690
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tosk, Inc. (Industry)
Collaborators: SIRO Clinpharm Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLP-2690-0007
Record Dates: First submitted 2022-12-05; First posted 2023-01-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Mucositis
Keywords: Mucositis; Uridine Phosphorylase Inhibitor; Chemotherapy; 5 FU/ LU; Colorectal cancer
MeSH Terms: conditions — Mucositis; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 24 patients will be enrolled into one of 2 different: TK112690 treated or placebo treated
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be partially blinded. The patient and investigator as well as site personnel will be blinded as to whether TK-90 or TK-90 placebo is administered. The CRO, sponsor, and site pharmacist will know whether the patient was administered active drug or TK-90 placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TK112690 (Experimental): TK112690 treatment
  Interventions: Drug: TK-112690
- Placebo (Placebo Comparator): TK112690 formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TK-112690 — TK112690 treatment Post 5-FU chemotherapy
  Arms: TK112690
Drug: Placebo — Placebo treatment Post 5-FU chemotherapy
  Arms: Placebo

SUMMARY:
Patients expected to receive a 500 mg/m2 of Leucovorin by iv & 500 mg/m2 of Fluorouracil (5FU) by iv bolus for their Colorectal Cancer. The patients will receive a one-hour infusion of TK-90 or equivalent TK-90 placebo depending on randomization at 5 hours & 11 hours post 5-FU iv bolus. This treatment cycle will continue weekly for 6 weeks. The TK112690 dose will be 45 mg/kg.

DETAILED DESCRIPTION:
Patients expected to receive a 500 mg/m2 of Leucovorin by iv & 500 mg/m2 of Fluorouracil (5FU) by iv bolus for their Colorectal Cancer. The patients will receive a one-hour infusion of TK-90 or equivalent TK-90 placebo depending on randomization at 5 hours & 11 hours post 5-FU iv bolus. This treatment cycle will continue weekly for 6 weeks. The TK112690 dose will be 45 mg/kg.

* 24 patients will be randomized equally into 2 different groups: TK-90 treated or TK-90 placebo treated.
* Screening must be completed within 2 weeks.
* The treatment period for the study is 6 weeks.
* Study follow-up will be scheduled post two weeks of completion of last dose of Chemotherapy & TK-90
* Blinding: The study will be partially blinded. The patient and investigator as well as site personnel will be blinded as to whether TK-90 or TK-90 placebo is administered. The CRO, sponsor, and site pharmacist will know whether the patient was administered active drug or TK-90 placebo

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 to 75 years old (both inclusive) with a histologically or cytological confirmed diagnosis of colorectal cancer
2. Patient scheduled to receive bolus 5 FU along with LV as first line or subsequent therapy for treating locally advanced or residual or recurrent or metastatic colorectal cancer.
3. No prior systemic treatments for cancer (chemotherapy and/or radiotherapy) 4 weeks prior to screening.
4. Be able to read and understand and provide a signature or thumb impression on the Informed Consent Form (ICF) before entering the study.
5. No other concurrent, active, invasive malignancy.
6. ECOG performance status of 0 to 2.
7. Must have a life expectancy of at least 6 months.
8. No active angina or uncontrolled arrhythmia.
9. Not pregnant or nursing. Women of childbearing potential must have a negative serum pregnancy test at screening and on the day before dosing and must use medically acceptable methods of birth control. Acceptable methods of birth control include oral or transdermal contraceptives, condoms, spermicidal foam, IUD, progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or post-menopausal for more than or equal to 1 year, must be specified in the patient's medical history file and CRF.
10. Mucositis Grade less than or equal to 1 per WHO Scale and Xerostomia of Grade less than or equal to 2 per CTCAE
11. Adequate bone marrow function as per CTCAE V5, defined as follows:

    i) Absolute neutrophil count more than or equal to 1500 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to randomization ii) Platelets more than or equal to 100,000 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to randomization iii) Hemoglobin more than or equal to 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to randomization (Note: The use of transfusion or other intervention to achieve Hgb more than 8.0 g/dl is acceptable).
12. Adequate hepatic function with bilirubin less than or equal to 1.5 x upper-normal limit (ULN), AST or ALT less than or equal to 3x ULN within 2 weeks prior to randomization
13. Adequate renal function with serum creatinine less than 1.5 mg/dl and creatinine clearance (CrC) more than or equal to 50 ml/min within 2 weeks prior to randomization determined by 24-hour collection or estimated by Cockcroft-Gault formula. CrC male is equal to [(140 - age) x (wt in kg)] / [(Serum Cr mg/dl) x (72)]. CrC female is equal to 0.85 x (CrCl male)
14. Normal serum calcium or normal corrected serum calcium within 2 weeks prior to randomization; formula for corrected calcium if albumin valued is below normal range: Corrected calcium (mg/dl) is equal to (4 - [patients albumin (g/dl)] x 0.8) + patient measured calcium (mg/dl).

Exclusion Criteria:

1. An active infection including HIV/ HBV/ HCV infection.
2. Patients who have not fully recovered after prior surgery. (Patients who have had prior surgery and have fully recovered and patients who may have surgery in the future are eligible.)
3. Unstabilized or symptomatic brain metastasis (History of brain metastases allowed if disease has stabilized or improved after radiation and/or craniotomy).
4. Pregnant or nursing mother.
5. Prior history of a cerebrovascular accident or hemorrhage.
6. Congestive heart failure, as defined by New York Heart Association class III or IV.
7. Uncontrolled hypertension.
8. Active psychiatric/mental illness making informed consent or useful clinical follow-up unlikely.
9. Patients who have previously been enrolled into this study and subsequently withdrew.
10. Patient receiving other investigational agent(s).
11. Any systemic immunosuppressive medication/therapy (eg, other chemotherapy, steroids).
12. Any prohibited prior or concomitant therapy 2 weeks prior to enrollment.
13. Presence of any significant systemic illness, unstable or severe medical condition(s) that could put the patient at risk during the study, interfere with outcome measures, or affect compliance with the protocol procedures such as intercurrent infection and/or autoimmune disease, ie, any condition that compromises the immune system.
14. Known or suspected intolerance or hypersensitivity to the study materials (TK 90 and/or excipients or closely related compounds).
15. Patients that have a history of poor compliance in clinical research studies.
16. Patients that have participated in any other investigative clinical trial in the past 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Mucositis | 8 Weeks
  SOM (Severe Oral Mucositis) - Comparison of incidences of Grade 3 or 4 mucositis (WHO scale) in the treatment and placebo groups.
  Duration of SOM. Days patients suffer Grades 3 and 4 oral mucositis measured by WHO scale from the start of treatment. number of days from the first occurrence of WHO Grade 3 or 4 OM through the first occurrence of non-severe (≤ Grade 2) without a subsequent instance of ≥ Grade 3 OM. Subjects with complete study follow-up for severe OM who do not develop severe OM (grade 0-2) will be considered to have durations of 0 days

SECONDARY OUTCOMES:
Secondary efficacy/outcome mucositis | 8 Weeks
  A) In addition to the WHO scale, mucositis status in the patients will also be evaluated using two different published and validated mucositis scales: NCI/CTCAE/mucositis, and PROMS.
  B) Comparison of WHO scale values of treated patients at each point of evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Emile Youssef, MD, PhD, Study Director — Tosk, Inc.
Locations (5):
- India (5):
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal, Madhya Pradesh
  - Om Sai Onco Surgery Multispecialty Hospital Center, Kolhāpur, Maharashtra
  - B. J. Medical College and Sassoon General Hospital, Pune, Maharashtra
  - MTES Sanjeevan Hospital, Pune, Maharashtra
  - Saveetha Medical college Chennai, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No